CLINICAL TRIAL: NCT05161923
Title: To Evaluate the Nutritional Parameters in Patients With Achalasia
Brief Title: COMPREHENSIVE ANALYSIS OF NUTRITIONAL PARAMETERS IN PATIENTS WITH IDIOPATHIC ACHALASIA: A PROSPECTIVE STUDY.
Acronym: POEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Clinical Professor, Asian Institute of Gastroenterology, India
Other Study IDs: HREM1
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Weight Gain; Nutritional Imbalance
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Per oral endoscopy myotomy: The per-oral endoscopic myotomy, or POEM, is a minimally invasive surgical procedure for the treatment of achalasia wherein the inner circular muscle layer of the lower esophageal sphincter is divided through a submucosal tunnel.[1] This enables food and liquids to pass into the stomach, a process that is impaired in achalasia. The tunnel is created, and the myotomy performed, using a flexible endoscope, meaning the entire procedure can be done without external incisions.
  Interventions: Procedure: Per oral endoscopy myotomy

INTERVENTIONS:
Procedure: Per oral endoscopy myotomy — The per-oral endoscopic myotomy, or POEM, is a minimally invasive surgical procedure for the treatment of achalasia wherein the inner circular muscle layer of the lower esophageal sphincter is divided through a submucosal tunnel.[1] This enables food and liquids to pass into the stomach, a process that is impaired in achalasia. The tunnel is created, and the myotomy performed, using a flexible endoscope, meaning the entire procedure can be done without external incisions.
  Other Names: POEM

SUMMARY:
A total of 100 patients aged 18-60 years with confirmed diagnosis of achalasia cardia will be recruited prospectively. In this study, patients diagnosed with achalasia cardia (prior to per oral endoscopic myotomy treatment) will undergo comprehensive evaluation of their nutritional status. All the participants will be asked about the details enlisted in pre-tested proforma.The evaluation will include demographic data(age, gender, food preferences, socio economic status,underlying diseases such as hypertension diabetes mellitus etc) anthropometric assessment (height, weight, Body Mass Index, weight loss and duration, percentage weight loss, midupperarm circumference , triceps skin fold, hand grip strength) and biochemical assessment (Hemoglobin, serum albumin and serum pre-albumin,total protein, serum Vitamin D, calcium, B12, serum iron). Each patients' dietary habits will be assessed by SUBJECTIVE GLOBAL ASSESMENT questionnaire (weight change, dietary intake, gastrointestinal symptoms, functional capacity, oedema, subcutaneous fat,muscle wasting, ascites.The obtained data will be statistically analyzed and interpreted. As we are in the midst of COVID-19 pandemic, we will be taking utmost safety precautions to prevent cross-infection. The doctor performing the study and the accompanying technician will be donning the personal protection equipment all throughout the study.

DETAILED DESCRIPTION:
1. .STUDY DESIGN: This study is a Prospective single arm observational study.
2. .STUDY PERIOD: Jan 2021-May 2021. 3. SAMPLE SIZE: 100 participants.

INCLUSION CRITERIA:

1. Male and female patients aged 18-60 years with confirmed diagnosis of idiopathic achalasia.
2. Patients who are co-operative, can communicate verbally and willing to give informed consent.

   EXCLUSION CRITERIA:
3. Chronic diarrhea, malignancy, severe comorbid illness affecting the nutritional status
4. Previously treated and asymptomatic cases with achalasia

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-60 years with confirmed diagnosis of idiopathic achalasia.
2. Patients who are co-operative, can communicate verbally and willing to give informed consent.

Exclusion Criteria:

1. Chronic diarrhea, malignancy, severe comorbid illness affecting the nutritional status
2. Previously treated and asymptomatic cases with achalasia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-12-25 (Estimated); Study Completion 2022-03-26 (Estimated)

PRIMARY OUTCOMES:
To assess the various nutritional indices in cases with treatment ( per oral endoscopic myotomy) failure cases with idiopathic achalasia | 12 months
  To assess the detailed biochemical assessment i.e., change in the levels of hemoglobin, serum albumin, total protein, vitamin D, calcium, vitamin B12 before and after the per oral endoscopic myotomy procedure.

SECONDARY OUTCOMES:
To evaluate the severity of malnutrition before and after undergoing Per-oral endoscopic myotomy (Per Oral Endoscopic Myotomy). | 12 months
  To determine the anthropometric assessment i.e., amount of weight loss or weight gain and its duration, change in triceps skinfold and midupperarm circumference of patients diagnosed with idiopathic achalasia.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MBBS MD DNB, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

REFERENCES:
- [Derived] Nabi Z, Basha J, Inavolu P, Goud R, Veligatla V, Tummuru SP, Cheripelli N, Arutla M, Ramchandani M, Darisetty S, Nageshwar Reddy D. Comprehensive analysis of nutritional parameters in patients with idiopathic achalasia: A prospective study in India. Indian J Gastroenterol. 2025 Feb;44(1):57-63. doi: 10.1007/s12664-024-01664-5. Epub 2024 Aug 19. PMID 39158832